CLINICAL TRIAL: NCT06899282
Title: The Effect of Pressure Ulcer Management Program Applied With Jigsaw Technique on Nursing Students' Pressure Ulcer Knowledge, Attitude and Self-efficacy: A Double-blind Randomized Controlled Trial
Brief Title: The Effect of Pressure Ulcer Management Program Applied With Jigsaw Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Senay Takmak, Assistant Professor, Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2025/03-13
Record Dates: First submitted 2025-03-17; First posted 2025-03-27 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Pressure Ulcers; Nursing Students; Training Effectiveness; Randomized Controlled Trial
Keywords: jigsaw technique; nursing student; training effectiveness; randomized controlled trial; pressure ulcers
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group: The group to be taught with jigsaw technique. (Experimental): Intervention Group: The lecture on pressure ulcer prevention and management to the intervention group will be conducted with the jigsaw technique. Pressure ulcer knowledge, attitude and prevention self-efficacy will be evaluated with standardized tools before, after the theoretical training and at the end of clinical practice. In addition, a standard student opinion questionnaire regarding the method will be applied.
  Interventions: Behavioral: Jigsaw method
- Control Group: This is the group that will receive theoretical training with the traditional method. (Active Comparator): Control group: Control group students will receive theoretical training prepared by the researchers. Pressure ulcer knowledge, attitude and prevention self-efficacy will be evaluated with standardized tools before, after the theoretical training and at the end of clinical practice.
  Interventions: Behavioral: The theoretical training

INTERVENTIONS:
Behavioral: Jigsaw method — Jigsaw/puzzle method is one of the collaborative learning techniques. The Jigsaw technique requires each student to focus on a particular aspect of the topic, become an "expert" on that topic and teach it to their peers. Once the students have learned the topic in their expert group, they return to the original group and teach what they have learned back to them as if solving a jigsaw puzzle (Geiselman et al., 2024). For the application of the technique, the "Jigsaw Technique Application Directive" was prepared as a training material to be delivered to the students.
  Arms: Intervention group: The group to be taught with jigsaw technique.
Behavioral: The theoretical training — The theoretical training will be conducted in 2 sessions. The first session will cover the definition, prevalence and importance of pressure ulcers, etiology and classification, risk assessment and pressure ulcers in special patient groups. The second session will cover prevention and treatment of pressure ulcers.
  Arms: Control Group: This is the group that will receive theoretical training with the traditional method.

SUMMARY:
The aim of this study is to evaluate the effectiveness of the jigsaw method on pressure ulcer prevention in senior nursing students. In addition, the study will also examine student views on the jigsaw technique.

Hypotheses of the study are as follows:

Hypothesis 1: The pressure injury management program applied with the Jigsaw technique has an effect on the pressure ulcer knowledge scores of nursing students.

Hypothesis 2: The pressure injury management program applied with the Jigsaw technique has an effect on the pressure ulcer prevention attitude of nursing students.

Hypothesis 3: The pressure injury management program applied with the Jigsaw technique has an effect on nursing students' pressure ulcer management self-efficacy.

The participant characteristics were being a 4th grade student of Kütahya University of Health Sciences, Faculty of Health Sciences, Department of Nursing and being enrolled in the Basic Principles and Practices in Nursing Practices Course. Nursing students who did not volunteer to participate in the study, those who did not participate in theoretical and clinical practices during the academic semester, and nursing students working as high school graduate nurses due to their past education will be excluded from the study.

Intervention and measurements: Participants (N=70) will be randomly divided into intervention and control groups. The intervention group will study pressure ulcer management with the jigsaw technique. The control group will receive theoretical education with the traditional method. Students' pressure ulcer knowledge, attitude and self-efficacy levels will be assessed with standardized tools. Baseline assessment before the intervention, post-intervention and 6 weeks after the intervention will be done. Measurements will be made by students through self-reporting. However, a researcher blinded to the groups will administer the instruments and enter data. Data analysis will also be done by the researcher blinded to the groups. Thus, double blindness will be ensured. Statistical analysis will be based on significance tests.

DETAILED DESCRIPTION:
Nurses should identify patients at high risk of pressure ulcers and provide preventive care accordingly. However, two recently published meta-analysis studies found that the pressure ulcer knowledge of nurses and nursing students measured by standard tools was below the acceptable level (60%). However, the attitudes of nursing students towards pressure ulcer prevention were found to be positive and at a high level. In addition, a multicentre study conducted in Türkiye showed that nursing students' self-efficacy in pressure ulcer prevention was also low and there was a positive relationship between knowledge and self-efficacy. This situation reveals the need for the use of better educational methods to improve nursing students' pressure ulcer knowledge.

Nursing educators are responsible for improving students' knowledge, skills and attitudes about pressure ulcers and preparing them for clinical practice. In the literature, there are studies showing that active teaching methods such as six-hat thinking technique, case-supported concept map, make significant improvements in some results including nursing students' pressure sore knowledge. However, no study evaluating the effect of jigsaw technique on nursing students' pressure ulcer knowledge, attitudes and self-efficacy has been found. A meta-analysis study examining the results of the jigsaw technique in nursing students reported that the technique was an effective method in the results of students such as knowledge, skills and attitudes. In this context, this study was planned to evaluate the effectiveness of the jigsaw method on pressure ulcer prevention in senior nursing students.

ELIGIBILITY:
Inclusion Criteria:

* To be a 4th year student of the Department of Nursing, Faculty of Health Sciences, Kütahya University of Health Sciences
* To be enrolled in the Basic Principles and Practices in Nursing Course

Exclusion Criteria:

* Nursing students who did not volunteer to participate in the study
* Not participating in theoretical and clinical practices during the academic semester
* Graduated from health vocational high school and working with the title of nurse

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2025-04-11 (Actual); Primary Completion 2025-06-06 (Actual); Study Completion 2025-06-06 (Actual)

PRIMARY OUTCOMES:
Pressure Ulcer Knowledge Assessment Tool-Updated Version | Baseline (Time 0), After 4 hours (Time 1), After 6 weeks (Time 2)
  Pressure Ulcer Knowledge Assessment Tool-Updated is a tool that measures nurses' knowledge about pressure ulcers within the framework of evidence-based guidelines.It consists of 25 multiple-choice questions on six themes: Etiology, Classification and Observation, Risk Assessment, Nutrition, Prevention of Pressure Ulcers and Specific Patient Groups. In scoring, 1 point is given for each correct answer and 0 points for incorrect and "Don't know" answers. The total score ranges from 0 to 25. Cronbach's alpha value is 0.72.
Pressure Ulcer Prevention Attitude Scale | Baseline (Time 0), After 4 hours (Time 1), After 6 weeks (Time 2)
  Pressure Ulcer Prevention Attitude Scale The scale aims to assess attitudes towards pressure ulcer prevention. It consists of 13 items and 5 subscales including personal competence to prevent pressure ulcers (3 items), priority of pressure ulcer prevention (3 items), impact of pressure ulcers (3 items), personal responsibility in pressure ulcer prevention (2 items) and confidence in the effectiveness of prevention (2 items). Seven items (items 3, 5, 7, 8, 9, 10 and 13) are reverse scored as they are negative. The items are scored on a 4-point Likert scale (1 = strongly disagree, 4 = strongly agree) and score between 13 and 52 points. A higher score is interpreted as a more positive attitude. The Cronbach's alpha values of the original scale and the Turkish adaptation study are 0.79 and 0.71, respectively.
Pressure Ulcer Management Self-Efficacy Scale for Nurses | Baseline (Time 0), After 4 hours (Time 1), After 6 weeks (Time 2)
  The scale measures nurses' self-efficacy in managing pressure ulcers. The scale consists of a total of 10 items and four main subscales: Assessment, Planning, Supervision and Decision Making. Each item is scored from 1 (not at all competent) to 5 (completely competent). The scale does not include reverse items. The total score range is 0-100. The level of self-efficacy increases with the total score. The Cronbach Alpha value of the scale is 0.83.

OTHER OUTCOMES:
Jigsaw Opinion Scale | After training (only intervention group after jigsaw technique)
  Jigsaw Opinion Scale was developed by Şimşek (2007). It provides an assessment of students' views on learning with the jigsaw technique. The scale has a structure in which positive/negative opinions are asked with 14 five-point Likert items and one open-ended question comparing the jigsaw technique with the traditional learning method. The scale is scored between 14-70, and an increase in score is interpreted as the jigsaw technique being more effective than the traditional method. The Cronbach alpha value of the scale was calculated as 0.83 (Şimşek, 2007).

CONTACTS AND LOCATIONS:
Overall Officials: Necibe Dağcan Şahin, Asst. Prof., Study Chair — Kutahya Health Science University; Ferzan Kalaycı Emek, RA, Study Chair — Kutahya Health Science University; Burcu Nal, Asst. Prof., Study Chair — Kutahya Health Science University
Locations (1):
- Kütahya Health Science Univercity, Kütahya, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Research data can be shared upon request from the authors.

REFERENCES:
- [Background] Turhan Damar H, Erkin O. The effect of case-supported concept map education on nursing students' knowledge of and attitudes toward pressure injury prevention. J Tissue Viability. 2025 Feb;34(1):100848. doi: 10.1016/j.jtv.2024.12.012. Epub 2024 Dec 9. PMID 39665940
- [Background] Ozkan S, Uslusoy ECN. Outcomes of jigsaw technique in nurse education: A systematic review and meta-analysis. Nurse Educ Pract. 2024 Feb;75:103902. doi: 10.1016/j.nepr.2024.103902. Epub 2024 Jan 20. PMID 38301377
- [Background] Dalli OE, Yildirim Y, Caliskan G, Girgin NK. Reliability and validity of the Turkish version of pressure ulcer knowledge assessment tool-updated version (PUKAT 2.0). J Tissue Viability. 2022 Feb;31(1):52-57. doi: 10.1016/j.jtv.2021.08.001. Epub 2021 Aug 11. PMID 34429220
- [Background] Iseri O, Ursavas FE. The influence of the online education provided using the six thinking hat method on the knowledge and attitudes of nursing students regarding pressure injury prevention; a pilot study. J Tissue Viability. 2024 Aug;33(3):465-471. doi: 10.1016/j.jtv.2024.04.009. Epub 2024 Apr 16. PMID 38679544